CLINICAL TRIAL: NCT00281281
Title: Pharmacokinetics and Posology of Vancomycin in Adults Receiving ECMO
Brief Title: Pharmacokinetics of Vancomycin in Adults Receiving ECMO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9461701147
Record Dates: First submitted 2006-01-22; First posted 2006-01-24 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Extracorporeal Membrane Oxygenation
Keywords: Extracorporeal Membrane Oxygenation; vancomycin
MeSH Terms: interventions — Vancomycin

INTERVENTIONS:
Drug: vancomycin

SUMMARY:
1. Vancomycin is a drug that requires precise dosing and close monitoring to avoid drug toxicity.
2. There is limited data on the change of vancomycin pharmacokinetics in patients who need extracorporeal membrane oxygenation (ECMO).
3. This control trial is to understand:

   1. whether the pharmacokinetics of vancomycin is influenced by the use ECMO
   2. design the most appropriate dose of vancomycin in adult patients using ECMO.

DETAILED DESCRIPTION:
1. Vancomycin is a drug that requires precise dosing and close monitoring to avoid drug toxicity.
2. Oftentimes it is used in intensive care units (ICU) for patients who need a life-saving machine for heart and lung failure called extracorporeal membrane oxygenation (ECMO).
3. There is limited data on the change of vancomycin pharmacokinetics in these patients.
4. This is a control trial using ICU patients who need vancomycin but not ECMO as a control to understand:

   1. whether the pharmacokinetics of vancomycin is influenced by the use ECMO
   2. design the most appropriate dose of vancomycin in adult patients using ECMO.
5. After the 4th dose of vancomycin, blood was drawn at appropriate time spots (1 mL each) to determine the time concentration curve and to calculate the pharmacokinetic parameters for 2 groups of patients to determine if there is any difference.

ELIGIBILITY:
Inclusion Criteria:

* >18 y/o
* receiving ECMO for study group
* without ECMO for control group (sex, age, creatinine clearance match with study group)

Exclusion Criteria:

* severe burn (>30-40% BSA)
* receiving continuous renal replacement therapy or hemodialysis concurrently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2005-12; Study Completion 2007-04

PRIMARY OUTCOMES:
pharmacokinetic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Fe-Lin L Wu, MSCP, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan